CLINICAL TRIAL: NCT00100880
Title: A Phase I Trial of CC-5013 (Lenalidomide) in Pediatric Patients With Recurrent or Refractory Primary CNS Tumors
Brief Title: Lenalidomide in Treating Young Patients With Recurrent, Progressive, or Refractory CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03176; NCI-2012-03176 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR653734; PBTC-018 (Other: Pediatric Brain Tumor Consortium); PBTC-018 (Other: CTEP); U01CA081457 (NIH); NCT00106990 (obsolete NCT alias)
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Childhood Atypical Teratoid/Rhabdoid Tumor; Childhood Central Nervous System Germ Cell Tumor; Childhood Choroid Plexus Tumor; Childhood Craniopharyngioma; Childhood Ependymoblastoma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood High-grade Cerebellar Astrocytoma; Childhood High-grade Cerebral Astrocytoma; Childhood Infratentorial Ependymoma; Childhood Low-grade Cerebellar Astrocytoma; Childhood Low-grade Cerebral Astrocytoma; Childhood Medulloepithelioma; Childhood Mixed Glioma; Childhood Oligodendroglioma; Childhood Supratentorial Ependymoma; Recurrent Childhood Brain Tumor; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma
MeSH Terms: conditions — Rhabdoid Tumor; Choroid Plexus Neoplasms; Astrocytoma; Oligodendroglioma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma | interventions — Lenalidomide

ARMS (1):
- Treatment (lenalidomide) (Experimental): Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 24 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 2-3 patients receive escalating doses of lenalidomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which an estimated 25% of patients experience dose-limiting toxicity.
  Interventions: Drug: lenalidomide; Procedure: perfusion-weighted magnetic resonance imaging; Procedure: diffusion-weighted magnetic resonance imaging; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Procedure: perfusion-weighted magnetic resonance imaging — Correlative studies
  Other Names: PW-MRI
Procedure: diffusion-weighted magnetic resonance imaging — Correlative studies
  Other Names: diffusion-weighted MRI
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of lenalidomide in treating young patients with recurrent, progressive, or refractory CNS tumors. Lenalidomide may stop the growth of CNS tumors by blocking blood flow to the tumor. It may also stimulate the immune system in different ways and stop tumor cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the MTD of oral CC-5013 administered to children with recurrent or refractory primary CNS tumors once daily for 21 days of a 28 day course.

II. To describe the toxicity profile and define the dose-limiting toxicity of CC-5013 in children with recurrent or refractory primary CNS tumors.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of CC-5013 in children and adolescents. II. To characterize the pharmacogenetics of CC-5013 in children and adolescents.

III. To evaluate changes in circulating endothelial cells (CECs) and circulating endothelial cell precursors (CEPs) in patients treated with CC-5013, and to investigate the correlation between changes in CECs and CEPs, plasma, serum and urine levels of proteins associated with angiogenesis including thrombospondin, b-FGF, TNF-α, IL-12, IL-8 and VEGF, and correlate these changes with changes in MR perfusion and clinical outcome.

IV. To evaluate changes in MR perfusion and diffusion during treatment.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 24 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 2-3 patients receive escalating doses of lenalidomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which an estimated 25% of patients experience dose-limiting toxicity.

All patients are followed for at least 30 days after the last dose of lenalidomide. Patients with treatment-related toxicity are followed for up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological diagnosis of a primary CNS tumor (including histologically benign brain tumors (e.g. low-grade glioma) that is recurrent, progressive, or refractory to standard therapy; patients with intrinsic brain stem or diffuse optic pathway tumors do not require histological confirmation of disease but should have clinical and/or radiographic evidence of progression
* Karnofsky Performance Scale (KPS for >= 16 yrs of age) or Lansky Performance Score (LPS for ≤ 16 years of age) ≥ 60 assessed within two weeks prior to registration
* Patient must be able to swallow capsules
* Patients must have recovered from any significant acute toxicity associated with prior therapy; patients must have no known curative therapy available; patients will be eligible regardless of the number of prior therapies, as long as other eligibility criteria are met
* Chemo: Prior use of thalidomide is acceptable; patients must have:

  * Received their last dose of known myelosuppressive anticancer chemotherapy or biological therapy at least three (3) weeks prior to study registration
  * Received their last dose of nitrosourea or mitomycin-C at least six (6) weeks prior to study registration
  * Received their last dose of other investigational agent or an anticancer drug known to not be myelosuppressive at least seven (7) days prior to study registration
* XRT: Patients must have had their last fraction of craniospinal irradiation ≥ 3 months prior to registration and their last fraction of local irradiation to primary tumor ≥ 4 weeks prior to registration
* Bone Marrow Transplant: ≥ 6 months since allogeneic bone marrow transplant and ≥ 3 months since autologous bone marrow/stem cell prior to registration
* Growth factors: Off all colony forming growth factor(s) > 2 weeks prior to registration (filgrastim, sargramostim, erythropoietin)
* The following laboratory values must be assessed within two (2) weeks prior to registration and again within seven (7) days prior to the start of therapy; laboratory tests should be repeated within 48 hours of beginning therapy if there has been a significant clinical change
* Absolute neutrophil count ≥ 1000/μl (unsupported)
* Platelets ≥ 100,000/μl (unsupported)
* Hemoglobin ≥ 8.0 g/dL (may be supported)
* Serum creatinine within upper limit of institutional normal for age
* Or GFR ≥ 70 ml/min/1.73m^2
* Bilirubin ≤ 1.5 times upper limit of normal for age
* SGPT (ALT) ≤ 2.5x institutional upper limit of normal for age
* Albumin ≥ 2 g/dL
* No overt renal, hepatic, cardiac or pulmonary disease
* Female patients of childbearing potential must have negative serum or urine pregnancy test (sensitivity of at least 50mIU/ml); patients must not be pregnant or breast-feeding
* All sexually active females must begin 2 methods of birth control, including 1 highly effective method, and 1 additional method (at the same time) at least 4 weeks prior to the first dose of CC-5013; this applies to all sexually active females of childbearing potential unless they have not had a menstrual period in 2 years or have undergone a hysterectomy
* Patients of child fathering potential must agree to use latex condoms during intercourse with a woman while taking CC-5013 and for 4 weeks thereafter
* Signed informed consent according to institutional guidelines must be obtained

Exclusion Criteria:

* Patients with a body surface area (BSA) ≤ 0.4 m^2 are excluded
* Patients with a first-degree relative with a history of venous thrombosis before age 50 yrs or an arterial thrombosis before age 40 yrs are excluded
* Patients who have had a thromboembolic event that is not line-related are excluded
* Patients with any significant medical illnesses that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise a patient's ability to tolerate this therapy
* Patients with any disease that would obscure toxicity or dangerously alter drug metabolism
* Patients receiving any other chemotherapeutics or investigational agents
* Patients with uncontrolled infection
* Patients unable to swallow capsules
* Patients with known hypersensitivity to anhydrous lactose, microcrystalline cellulose, croscarmellose sodium, and magnesium stearate

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2004-11; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
MTD, estimated using the modified Continual Reassessment Method (CRM) | 28 days

SECONDARY OUTCOMES:
Plasma drug concentrations and pharmacokinetic parameters, including volume of the central compartment (Vc/F), elimination rate constant (Ke), half-life (t1/2), apparent oral clearance (CL/F), and area under the plasma concentration time curve (AUC) | Baseline and course 1
  Presented in tabular and graphical form and determined using compartmental methods. Dose proportionality in pharmacokinetic parameters will be determined by performing one-way analysis of variance (ANOVA) on dose-normalized parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Warren, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (1):
- Pediatric Brain Tumor Consortium, Memphis, Tennessee, United States